CLINICAL TRIAL: NCT05507593
Title: A Multicenter Phase I Trial on the Safety and Preliminary Efficacy of DLL3-CAR-NK Cells in the Treatment of Relapsed / Refractory Extensive Stage Small Cell Lung Cancer
Brief Title: Study of DLL3-CAR-NK Cells in the Treatment of Extensive Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E20220808
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: SCLC, Extensive Stage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Patients of group A will be received 1x10^7 DLL3-CAR-NK cells infusion treatment.
  Interventions: Biological: DLL3-CAR-NK cells
- Group B (Experimental): Patients of group B will be received 1x10^8 DLL3-CAR-NK cells infusion treatment.
  Interventions: Biological: DLL3-CAR-NK cells
- Group C (Experimental): Patients of group C will be received 1x10^9 DLL3-CAR-NK cells infusion treatment.
  Interventions: Biological: DLL3-CAR-NK cells

INTERVENTIONS:
Biological: DLL3-CAR-NK cells — Patients of Group A will be received 1x10^7 DLL3-CAR-NK cells infusion treatment，of group B will be received 1x10^8 DLL3-CAR-NK cells infusion treatment，and of group C will be received 1x10^9 DLL3-CAR-NK cells infusion treatment.

SUMMARY:
This is a multicenter, open-label, phase I clinical trial aimed to evaluate the safety and efficacy of DLL3-CAR-NK cells treatment for relapsed and refractory extensive small cell lung cancer (ES-SCLC).

DETAILED DESCRIPTION:
This study is a multicenter, single arm, open-label, non randomized, single dose, dose escalation, phase I clinical trial on relapsed and refractory ES-SCLC. The phase I clinical trial will be conducted according to the principle of "3 + 3". Three dose groups will be set up, namely group A: 1.0 × 10^7, group B: 1.0 × 10^8, and group C: 1.0 × 10^9 DLL3-CAR-NK cells. 9-18 subjects will be enrolled in the groups and given a single infusion of DLL3-CAR-NK cells injection in order to determine the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD), evaluate the safety and efficacy of the cell infusion. It well be recommend dose for phase II clinical study (recommended phase II dose, RP2D).

ELIGIBILITY:
Inclusion Criteria:

Only patient who meet all the following conditions can be selected for this trial:

1. Patients voluntarily sign informed consent;
2. The age was 18-75 years old, and the gender was not limited;
3. Patients who meet the following diagnosis and treatment : 1) small cell lung cancer diagnosed by tissue / cytology; 2) extensive small cell lung cancer diagnosed by imaging according to VALG and AJCC-8; 3) disease progression after receiving at least one line treatment, and disease progression within 6 months after the last line treatment;
4. The expected survival time was more than 3 months;
5. There are measurable target lesions on imaging during screening: the maximum diameter is greater than 1.0 cm;
6. The Eastern Cooperative Oncology Group (ECOG) scored 0 or 1 for physical fitness;
7. Sufficient bone marrow reserve at screening, defined as:

   * Neutrophil absolute value (ANC) > 1.5 × 10^9/L；
   * Lymphocyte absolute value (ALC) ≥ 0.3 × 10^9/L；
   * Platelet (PLT) ≥ 100 × 10^9/L；
   * Hemoglobin (HGB) ≥ 100g / L;
8. The screening has appropriate organ function and meets the following criteria:

   * Aspartate aminotransferase (AST) ≤ 2.5 times ULN (due to tumor infiltration ≤ 5 times ULN);
   * Alanine aminotransferase (ALT) ≤ 2.5 times ULN (due to tumor infiltration ≤ 5 times ULN);
   * Total serum bilirubin ≤ 1.5 times ULN (due to tumor infiltration ≤ 3 times ULN);
   * Serum creatinine (SCR) ≤ 1.5 times ULN, or creatinine clearance rate ≥ 60ml / min;
   * Have the lowest level of lung reserve, defined as ≤ grade 1 dyspnea and oxygen saturation > 91% in non oxygen breathing state;
   * International normalized ratio (INR) ≤ 1.5 times ULN, and activated partial prothrombin time (APTT) ≤ 1.5 times ULN;
9. Blood vessel conditions for collection of mononuclear cells are available during screening;
10. The urine pregnancy test of women of childbearing age is negative. Any male and female patient with fertility must agree to use effective contraceptive methods during the whole study and at least 1 year after the study treatment.

Exclusion Criteria:

Patient who meet any of the following conditions well excluded in this trial:

1. At the time of screening, patients with symptomatic central nervous system (CNS) metastases (asymptomatic CNS metastases, or asymptomatic after local treatment and stable condition for 4 weeks can be enrolled);
2. Those with a history of central nervous system before screening, such as epilepsy, cerebral ischemia / hemorrhage, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, cerebral organic syndrome, mental disease or any autoimmune disease involving the central nervous system;
3. Those who had received immunotherapy, targeted therapy, chemotherapy, or radiotherapy within 4 weeks before screening and were assessed by the investigator as unsuitable for inclusion;
4. Those who stopped systemic hormone therapy for less than 72 hours before cell transfusion; But it is allowed to use a physiological substitute amount of hormone (such as prednisone < 10mg / D or equivalent);
5. Those who have used any adoptive cell therapy before screening;
6. Those who have received organ / tissue transplantation before screening;
7. Active systemic autoimmune disease is known before screening and is under treatment;
8. Those who meet any of the following conditions during screening:

   * positive for hepatitis B surface antigen (HBsAg) and / or hepatitis B e antigen (HBeAg);
   * hepatitis B e antibody (HBE AB) and / or hepatitis B core antibody (HBC AB) are positive, and the copy number of HBV-DNA is greater than the lower measurable limit;
   * positive for hepatitis C antibody (HCV AB);
   * positive anti Treponema pallidum antibody (TP AB);
   * HIV antibody test positive;
   * the copy number of EBV-DNA and cmv-dna is greater than the lower measurable limit;
9. Those who had undergone major surgery within 4 weeks before screening and were assessed by the investigator as unsuitable for inclusion;
10. Those who had or were suffering from other malignant tumors within 2 years before screening;
11. The heart meets any of the following conditions during screening:

    * left ventricular ejection fraction (LVEF) ≤ 50% (echo);
    * New York Heart Association (NYHA) class III or IV congestive heart failure;
    * hypertension (systolic blood pressure ≥ 140mmHg and / or diastolic blood pressure ≥ 90mmHg) or pulmonary hypertension that has not been controlled by standard treatment;
    * have had myocardial infarction or cardiac surgery within 12 months before cell transfusion;
    * clinically significant valvular disease.
12. The tumors involved atrium or ventricle during screening;
13. Patients with history of pulmonary interstitial fibrosis or severe COPD;
14. There are clinical emergencies (such as intestinal obstruction or vascular compression) requiring urgent treatment due to tumor body obstruction or compression during screening;
15. Patients with active bleeding during screening;
16. Patients with deep venous thrombosis or pulmonary embolism within 6 months before screening;
17. Those who received live vaccine within 6 weeks before screening;
18. Patients with active infection and need treatment during screening;
19. Participated in other intervention clinical studies within 4 weeks before screening;
20. Poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
The dose-limiting toxicity (DLT) | 1 year
Maximum tolerated dose (MTD) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dingzhi Huang, M.D, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China